CLINICAL TRIAL: NCT06893913
Title: Effect of Addition of Pyramidal Exercise to Intermittent Fasting on Dryness of Eye in Pre-diabetic Psoriasis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, Department of Physical Therapy for Cardiovascular/Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004789
Record Dates: First submitted 2025-03-13; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis; PreDiabetes; Obesity; Dry Eye
MeSH Terms: conditions — Psoriasis; Prediabetic State; Obesity; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercised group (Experimental): twenty obese patients with dryness of eye, obesity, (prediabetes), and psoriasis will receive intermittent fasting consisted of eating ad libitum for 5 days and then will restrict calories ('fasting') for two days weekly, for 12 weeks. On the fasting days, participants will restrict calories to a maximum of 600 kcal/day for females and 650 kcal/day for males.
  The dietary intervention will be based on the 5:2 fasting diet. Subjects will be asked to consume a total of allowed calories in a window of 6 hours or less from 8:00 am till 2:00 pm, twice per week on 2 non-consecutive days.
  also this group will receive a pyramidal training nearly 60 minutes (nearly two rounds of 21 minutes of running on treadmill will be separated with 10 min of rest between the two rounds. Also, warming (4 min before start of pyrimidal trianing) and cooling (4 minu after pyramidal training) will be done through gentle stretching. the exercise will be applied 3 times weekly for 12 weeks
  Interventions: Behavioral: pyramidal training plus intermittent fasting
- non-exercised group (Active Comparator): twenty obese patients with dryness of eye, obesity, insulin resistance (prediabetes), and psoriasis (chronic plaque) will receive The intermittent fasting regimen consisted of eating ad libitum for five days and then will restrict calories ('fasting') for two days per week, for a duration of 12 weeks. On the fasting days, participants will be instructed to restrict their calories to a maximum of 600 kcal/day for females and 650 kcal/day for males.
  The intermittent fasting intervention will consist of a dietary intervention based on the 5:2 fasting diet. Subjects will be asked to consume a total of allowed calories in a window of 6 hours or less from 8:00 am till 2:00 pm, twice per week on 2 non-consecutive days.
  Interventions: Behavioral: intermittent fasting

INTERVENTIONS:
Behavioral: pyramidal training plus intermittent fasting — twenty obese patients with dryness of eye, obesity, (prediabetes), and psoriasis will receive intermittent fasting consisted of eating ad libitum for 5 days and then will restrict calories ('fasting') for two days weekly, for 12 weeks. On the fasting days, participants will restrict calories to a maximum of 600 kcal/day for females and 650 kcal/day for males.
  The dietary intervention will be based on the 5:2 fasting diet. Subjects will be asked to consume a total of allowed calories in a window of 6 hours or less from 8:00 am till 2:00 pm, twice per week on 2 non-consecutive days.
  also this group will receive a pyramidal training nearly 60 minutes (nearly two rounds of 21 minutes of running on treadmill will be separated with 10 min of rest between the two rounds. Also, warming (4 min before start of pyrimidal trianing) and cooling (4 minu after pyramidal training) will be done through gentle stretching. the exercise will be applied 3 times weekly for 12 weeks
  Arms: exercised group
Behavioral: intermittent fasting — twenty obese patients with dryness of eye, obesity, (prediabetes), and psoriasis will receive intermittent fasting consisted of eating ad libitum for 5 days and then will restrict calories ('fasting') for two days weekly, for 12 weeks. On the fasting days, participants will restrict calories to a maximum of 600 kcal/day for females and 650 kcal/day for males.
  The dietary intervention will be based on the 5:2 fasting diet. Subjects will be asked to consume a total of allowed calories in a window of 6 hours or less from 8:00 am till 2:00 pm, twice per week on 2 non-consecutive days.
  Arms: non-exercised group

SUMMARY:
insulin resistant psoriatic obese patients may complain problems of dryness of eye. Intermittent fasting may improve dryness of eye, obesity, insulin resistance, and psoriasis. Exercise, as applied in pyramidal form, if added to intermittent fasting may improve effect of intermittent fasting.

DETAILED DESCRIPTION:
forty obese patients with dryness of eye, obesity, insulin resistance (prediabetes), and psoriasis (chronic plaque) will randomly distributed to group I (n =20 patients) or group II (n=20). Both groups will receive The intermittent fasting regimen consisted of eating ad libitum for five days and then will restrict calories ('fasting') for two days per week, for a duration of 12 weeks. On the fasting days, participants will be instructed to restrict their calories to a maximum of 600 kcal/day for females and 650 kcal/day for males.

The intermittent fasting intervention will consist of a dietary intervention based on the 5:2 fasting diet. Subjects will be asked to consume a total of allowed calories in a window of 6 hours or less from 8:00 am till 2:00 pm, twice per week on 2 non-consecutive days.

Group I will receive a pyramidal training will be adopted for nearly 60 minutes (nearly two rounds of 21 minutes of running on electronic treadmill will be separated with 10 minutes of rest between the two rounds. Also, warming (4 minutes before start of pyrimidal trianing) and cooling (4 minutes after pyramidal training) will be done through gentle stretching exercises/activities. the exercise will be applied 3 times weekly for 2 weeks

ELIGIBILITY:
Inclusion Criteria:

* chronic plaque psoriasis
* obesity class I
* prediabetic persons
* dryness of both eyes

Exclusion Criteria:

* cardiac insults
* respiratory insults
* diabetics hypertensives or renal, hepatic insults

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
schrimer test | it will be assessed after 12 weeks
  it is a test for eye dryness

SECONDARY OUTCOMES:
Tear film break-up timing | it will be assessed after 12 weeks
  it is a test for eye dryness
System of Dry eye scoring | it will be assessed after 12 weeks
  it is a questionnaire for eye dryness assessment
Ocular surface disability index | it will be assessed after 12 weeks
  it is a questionnaire for eye dryness assessment
Dermatology life quality index | it will be assessed after 12 weeks
  it is a questionnaire for psoriasis-associated life quality assessment
Psoriasis area and severity index | it will be assessed after 12 weeks
  A PASI score is a tool used to measure the severity and extent of psoriasis. PASI is an acronym for Psoriasis Area and Severity Index.The PASI is a widely used instrument in psoriasis trials that assesses and grades the severity of psoriatic lesions. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease).
Fasting serum blood glucose | it will be assessed after 12 weeks
  it will measure of blood fasting glucose
Waist circumference | it will be assessed after 12 weeks
  it will be assessed via tape
Body mass index | it will be assessed after 12 weeks
  it will be assessed on empty stomach

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of physical therapy, Giza, Dokki, Egypt